CLINICAL TRIAL: NCT03376529
Title: A Single-center, Multi-arm, Open-label, Randomized, 3-period, Crossover, Phase 1 Study to Evaluate the DDI, PK, Safety, and Tolerability of Single Doses of SPR741 Co-administered With Three Different Antibiotics in Healthy Volunteers
Brief Title: Phase 1 Study to Evaluate DDI, PK, Safety, Tolerability of SPR741
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spero Therapeutics (Industry)
Collaborators: Simbec Research (Industry); QPS Holdings LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SPR741-102
Record Dates: First submitted 2017-12-05; First posted 2017-12-18 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Healthy Volunteers
Keywords: safety; tolerability; pharmacokinetics; drug-drug interaction; SPR741; antibiotic
MeSH Terms: interventions — SPR741; Ceftazidime; Piperacillin, Tazobactam Drug Combination; Aztreonam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SPR741/Ceftazidime (N=9) (Experimental): Nine (9) participants will be enrolled and assigned to receive SPR741 400 mg IV over 1 hour, SPR741 400 mg IV over 1 hour + ceftazidime1.0 gram IV over 1 hour, and ceftazidime 1.0 gram IV over 1 hour in a randomized sequence. One treatment will be administered during each of 3 dose periods within the assigned treatment arm.
  Interventions: Drug: SPR741; Drug: Ceftazidime
- SPR741/Piperacillin/tazobactam (N=9) (Experimental): Nine (9) participants will be enrolled and assigned to receive SPR741 400 mg IV over 1 hour, SPR741 400 mg IV over 1 hour + piperacillin/tazobactam 4.5 grams IV over 1 hour, and piperacillin/tazobactam 4.5 grams IV over 1 hour in a randomized sequence. One treatment will be administered during each of 3 dose periods within the assigned treatment arm.
  Interventions: Drug: SPR741; Drug: Piperacillin/tazobactam
- SPR741/Aztreonam (N=9) (Experimental): Nine (9) participants will be enrolled and assigned to receive SPR741 400 mg IV over 1 hour, SPR741 400 mg IV over 1 hour + aztreonam 1.0 gram IV over 1 hour, and aztreonam 1.0 gram IV over 1 hour in a randomized sequence. One treatment will be administered during each of 3 dose periods within the assigned treatment arm.
  Interventions: Drug: SPR741; Drug: Aztreonam

INTERVENTIONS:
Drug: SPR741 — 400 mg IV over 1 hour
Drug: Ceftazidime — 1.0 gram IV over 1 hour
  Arms: SPR741/Ceftazidime (N=9)
Drug: Piperacillin/tazobactam — 4.5 grams IV over 1 hour
  Arms: SPR741/Piperacillin/tazobactam (N=9)
Drug: Aztreonam — 1.0 gram IV over 1 hour
  Arms: SPR741/Aztreonam (N=9)

SUMMARY:
This is a Phase 1, single-center, multi-arm, open-label, randomized, three-period, crossover study to evaluate the drug-drug interaction, pharmacokinetics, safety, and tolerability of a single dose of SPR741 combined with each of 3 different partner antibiotics (ceftazidime or piperacillin/tazobactam or aztreonam) in healthy volunteers. Participants will be administered single doses of SPR741 alone, a single dose of SPR741 in combination with 1 of 3 different partner antibiotics, and the partner antibiotic alone in a randomized sequence. Twenty-seven (27) adult male and female normal healthy participants 18 to 55 years of age are planned to participate in the study. Women of childbearing potential will not be eligible to participate.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, multi-arm, open-label, randomized, three-period crossover study to evaluate the drug-drug interaction, pharmacokinetics, safety, and tolerability of a single dose of SPR741 combined with each of 3 different partner antibiotics (ceftazidime, piperacillin/tazobactam, and aztreonam) in healthy volunteers. Participants will be administered a single dose of SPR741 alone, a single dose of SPR741 in combination with 1 of the 3 different partner antibiotics, and a single dose of the partner antibiotic alone in a randomized sequence. Twenty-seven (27) adult male and female normal healthy participants 18 to 55 years of age are planned to participate in the study. Women of childbearing potential will not be eligible to participate. The study will consist of 3 phases: a screening phase, a treatment phase, and a follow-up phase.

The 3 treatment arms will be enrolled and dosed in parallel or in a staggered manner, as needed for scheduling.

All participants in the study will be monitored for safety after administration of the last dose of investigational product.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males and/or females (of non-childbearing potential), 18 to 55 years of age (inclusive) at the time of screening;
2. BMI ≥ 18.5 and ≤ 29.9 (kg/m2) and weight between 55.0 and 100.0 kg (inclusive);
3. Medically healthy without clinically significant abnormalities at the screening visit or Day -1, including:

   1. Physical examination, vital signs. Vital signs include temperature, heart rate, respiratory rate, and blood pressure;
   2. Triplicate ECGs taken at least 1 minute apart with QTcF interval duration less than 450 msec obtained as an average from the triplicate screening and pre-dose Day 1 ECGs after at least 5 min in a semi-supine quiet rest;
   3. Hemoglobin/hematocrit, white blood cell (WBC) count, and platelet count equal to or greater than the lower limit of normal range of the reference laboratory;
   4. Creatinine, BUN, ALT and AST equal to or less than the upper limit of normal for the reference laboratory; results of all other clinical chemistry and urine analytes without any clinically significant abnormality.

   Discussion between the PI and the Medical Monitor (MM) is encouraged regarding the potential significance of any laboratory value that is outside of the normal range during the pre-dose period.
4. Be non-smokers (including tobacco, e-cigarettes or marijuana) for at least 1 month prior to participation in the study;
5. Willing and able to provide written informed consent;
6. Be willing and able to comply with all study assessments and adhere to the protocol schedule;
7. Have suitable venous access for drug administration and blood sampling;
8. If female, be of non-childbearing potential (e.g. post-menopausal as demonstrated by FSH or surgical sterilization i.e., tubal ligation or hysterectomy). Provision of documentation is not required for female sterilization, verbal confirmation is adequate;
9. If male, a willingness not to donate sperm and if engaging in sexual intercourse with a female partner who could become pregnant, a willingness to use a condom in addition to having the female partner use a highly effective method of birth control (such as an intrauterine device, diaphragm, oral contraceptives, injectable progesterone, subdermal implants, or a tubal ligation). This criterion applies to males (and/or female partners) who are surgically sterile and must be followed from the time of first study drug administration until 90 days after the final administration of study drug.

Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic or neurological disease, including any acute illness or surgery within the past 3 months determined by the PI to be clinically relevant;
2. History of known or suspected Clostridium difficile infection;
3. History of seizure disorders;
4. Positive urine drug/alcohol testing at screening or check-in (Day -1);
5. Positive testing for HIV, HBsAg or HCV;
6. History of substance abuse or alcohol abuse (defined as those who consume more than 14 units of alcohol per week, and where this consumption is spread over less than 3 days, or those who regularly (weekly) consumed excessive amounts of alcohol (>8 units for men and >6 units for women in one consumption, excessive amounts as defined by the UK National Office of Statistics) within the previous 5 years;
7. Use of any prescription medication or any over-the-counter medication, herbal products, vitamins, diet aids or hormone supplements within 7 days prior to randomisation;
8. Documented hypersensitivity reaction or anaphylaxis to any medication;
9. Donation of blood or plasma within 30 days prior to randomisation, or loss of whole blood of more than 500 mL within 30 days prior to randomisation, or receipt of a blood transfusion within 1 year of study enrollment;
10. Participation in a New Chemical Entity clinical study within the previous 3 months or a marketed drug clinical study within the 30 days before the first dose of IMP. (Washout period between studies is defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study).
11. Any other condition or prior therapy, which, in the opinion of the PI, would make the volunteer unsuitable for this study, including unable to cooperate fully with the requirements of the study protocol or likely to be non-compliant with any study requirements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Maximum concentration (Cmax) | Days 1 to 2, Days 4 to 5, Days 7 to 8
  Blood draws will be taken pre-dose (within 10 minutes), 30 minutes following the start of infusion, end of infusion and at 75, 90, 105, and 120 minutes, 4, 8, 12, and 24 hours following start of infusion.
Pharmacokinetics: Area under the concentration-time curve from time 0 to last measurable time-point (AUC0-t) | Days 1 to 2, Days 4 to 5, Days 7 to 8
  Blood draws will be taken pre-dose (within 10 minutes), 30 minutes following the start of infusion, end of infusion and at 75, 90, 105, and 120 minutes, 4, 8, 12, and 24 hours following start of infusion.
Pharmacokinetics: Area under the concentration-time curve from time 0 to infinity (AUC0-inf) | Days 1 to 2, Days 4 to 5, Days 7 to 8
  Blood draws will be taken pre-dose (within 10 minutes), 30 minutes following the start of infusion, end of infusion and at 75, 90, 105, and 120 minutes, 4, 8, 12, and 24 hours following start of infusion.
Pharmacokinetics: Time to maximum concentration (Tmax) | Days 1 to 2, Days 4 to 5, Days 7 to 8
  Blood draws will be taken pre-dose (within 10 minutes), 30 minutes following the start of infusion, end of infusion and at 75, 90, 105, and 120 minutes, 4, 8, 12, and 24 hours following start of infusion.
Pharmacokinetics: Terminal Elimination Rate Constant (kel) | Days 1 to 2, Days 4 to 5, Days 7 to 8
  Blood draws will be taken pre-dose (within 10 minutes), 30 minutes following the start of infusion, end of infusion and at 75, 90, 105, and 120 minutes, 4, 8, 12, and 24 hours following start of infusion.
Pharmacokinetics: Terminal half-life (t1/2) | Days 1 to 2, Days 4 to 5, Days 7 to 8
  Blood draws will be taken pre-dose (within 10 minutes), 30 minutes following the start of infusion, end of infusion and at 75, 90, 105, and 120 minutes, 4, 8, 12, and 24 hours following start of infusion.
Pharmacokinetics: Terminal clearance (CL) | Days 1 to 2, Days 4 to 5, Days 7 to 8
  Blood draws will be taken pre-dose (within 10 minutes), 30 minutes following the start of infusion, end of infusion and at 75, 90, 105, and 120 minutes, 4, 8, 12, and 24 hours following start of infusion.
Pharmacokinetics: Volume of distribution (Vd) | Days 1 to 2, Days 4 to 5, Days 7 to 8
  Blood draws will be taken pre-dose (within 10 minutes), 30 minutes following the start of infusion, end of infusion and at 75, 90, 105, and 120 minutes, 4, 8, 12, and 24 hours following start of infusion.

SECONDARY OUTCOMES:
Safety measures: adverse events (AEs) | Day -1 to Day 9
  The types and frequency of AEs
Safety measures: Summary of type and frequency of concomitant medication | Day -1 to Day 9
  The type and frequency of medications used will be summarized
Safety measures: change in temperature (C/F) | Day -1 to Day 9
  Change from baseline to end of study
Safety measures: change in blood pressure (mmHg) | Day -1 to Day 9
  Change from baseline to end of study
Safety measures: change in heart rate (beats per minute) | Day -1 to Day 9
  Change from baseline to end of study
Safety measures: abnormal, clinically significant physical exam findings | Day -1 to Day 9
  Change from baseline to end of study
Safety measures: abnormal, clinically significant changes in electrocardiogram parameter (RR Interval) | Day -1 to Day 9
  Change from baseline to end of study
Safety measures: abnormal, clinically significant changes in electrocardiogram parameter (P wave) | Day -1 to Day 9
  Change from baseline to end of study
Safety measures: abnormal, clinically significant changes in electrocardiogram parameter (PR Interval) | Day -1 to Day 9
  Change from baseline to end of study
Safety measures: abnormal, clinically significant changes in electrocardiogram parameter (QRS) | Day -1 to Day 9
  Change from baseline to end of study
Safety measures: abnormal, clinically significant changes in electrocardiogram parameter (ST Segment) | Day -1 to Day 9
  Change from baseline to end of study
Safety measures: abnormal, clinically significant changes in electrocardiogram parameter (T Wave) | Day -1 to Day 9
  Change from baseline to end of study
Safety measures:abnormal, clinically significant changes in urinalysis from baseline to end of study | Day -1 to Day 9
  Change from baseline to end of study
Safety measures: abnormal, clinically significant hematology changes from baseline to end of study | Day -1 to Day 9
  Change from baseline to end of study
Safety measures: abnormal, clinically significant serum chemistry changes from baseline to end of study | Day -1 to Day 9
  Change from baseline to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Annelize Koch, MBChB, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research, Ltd., Merthyr Tydfil, Mid Glamorgan, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eckburg PB, Lister T, Walpole S, Keutzer T, Utley L, Tomayko J, Kopp E, Farinola N, Coleman S. Safety, Tolerability, Pharmacokinetics, and Drug Interaction Potential of SPR741, an Intravenous Potentiator, after Single and Multiple Ascending Doses and When Combined with beta-Lactam Antibiotics in Healthy Subjects. Antimicrob Agents Chemother. 2019 Aug 23;63(9):e00892-19. doi: 10.1128/AAC.00892-19. Print 2019 Sep. PMID 31262767